CLINICAL TRIAL: NCT00459693
Title: PET Evaluation of Brain Peripheral Benzodiazepine Receptors Using (11C)PBR28 in HIV-Seropositive Patients With (MCMD)
Brief Title: PET Evaluation of Brain Peripheral Benzodiazepine Receptors Using [11C]PBR28 in HIV-Seropositive Patients With (MCMD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 070129; 07-M-0129
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2014-08-28

CONDITIONS: HIV-Dementia; HIV-Associated Cognitive Motor Complex; AIDS Encephalopathy; AIDS Dementia Complex; AIDS-Related Dementia Complex; HIV Infections; Healthy
Keywords: HIV-Dementia; Brain; PET; PBR28; MCMD; HIV Positive; HIV Dementia; AIDS Related Dementia; Minor Cognitive Motor Disorder; Healthy Volunteer; HV
MeSH Terms: conditions — AIDS Dementia Complex; HIV Infections; HIV Seropositivity | interventions — (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine

INTERVENTIONS:
Drug: [11C]PBR28

SUMMARY:
The purpose of this protocol is to measure a receptor in the brain using positron emission tomography (PET) that is involved in inflammation.

DETAILED DESCRIPTION:
The peripheral benzodiazepine receptor (PBR) is distinct from central benzodiazepine receptors associated with GABAa receptors. Although PBR was initially identified in peripheral organs such as kidneys, endocrine glands and lungs, later studies identified PBR in the central nervous system. In normal conditions, PBR is expressed in low levels in some neurons and glial cells. PBR can be a clinically useful marker to detect neuroinflammation, because activated microglial cells in inflammatory areas express much greater levels of PBR than in microglial cells in resting conditions.

PBR has been imaged with positron emission tomography (PET) using [11C]1-(2-chlorophenyl-N-methylpropyl)-3-isoquinoline carboxamide (PK11195). However, this classical ligand provides low levels of specific signal. Recently we developed a new ligand, N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine [11C]PBR28, which showed much greater specific signal than [11C]PK11195 in non-human primates. ln the present protocol we plan to perform a kinetic brain imaging study with [11C]PBR28 in HlV-seronegative controls, HIV-seropositive, non-impaired patients, and HlV-seropositive patients with minor cognitive motor disorder(MCMD). Each subject will recieve a brain-dedicated PET scan with 20 mCi[(11)C]PBR28.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria (healthy control subjects) aged 18 50 years with history/physical exam, ECG, and laboratory tests, plus inclusion criteria listed will be included in the protocol.

1. HIV-seropositive based on ELISA and Western blot (except the HIV-seronegative subjects, who will have ELISA screening).
2. Capable of providing informed consent.
3. Ambulatory at initial visit.
4. If cognitively impaired, the degree of impairment will be MCMD, and not frank HIV-associated dementia.

EXCLUSION CRITERIA:

1. Current psychiatric illness or severe systemic disease based on history and physical exam
2. Current dependence on alcohol or substances other than nicotine.
3. Laboratory results from blood or urine tests that show clinically significant abnormalities.
4. Previous radiation exposure (X-rays, PET scans etc.) that would exceed research limits.
5. Pregnancy and breast feeding.
6. A history of brain disease.
7. Cannot lie on your back for long periods since the pictures will be taken for about 2.5 hours during which time you will have to lie still on the scanner bed.
8. More than moderate hypertension.
9. Positive result on urine screen for illicit drugs.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04-09; Primary Completion 2014-04-06 (Actual); Study Completion 2014-04-06 (Actual)

PRIMARY OUTCOMES:
Brain uptake of [11C]PBR28 (measured as distribution volume). | One brain PET scan in one outpatient visit to NIH per subject.

CONTACTS AND LOCATIONS:
Overall Officials: William C Kreisl, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anderson E, Zink W, Xiong H, Gendelman HE. HIV-1-associated dementia: a metabolic encephalopathy perpetrated by virus-infected and immune-competent mononuclear phagocytes. J Acquir Immune Defic Syndr. 2002 Oct 1;31 Suppl 2:S43-54. doi: 10.1097/00126334-200210012-00004. PMID 12394782
- [Background] Anholt RR, De Souza EB, Oster-Granite ML, Snyder SH. Peripheral-type benzodiazepine receptors: autoradiographic localization in whole-body sections of neonatal rats. J Pharmacol Exp Ther. 1985 May;233(2):517-26. PMID 2987488
- [Background] Amodio P, Wenin H, Del Piccolo F, Mapelli D, Montagnese S, Pellegrini A, Musto C, Gatta A, Umilta C. Variability of trail making test, symbol digit test and line trait test in normal people. A normative study taking into account age-dependent decline and sociobiological variables. Aging Clin Exp Res. 2002 Apr;14(2):117-31. doi: 10.1007/BF03324425. PMID 12092785